CLINICAL TRIAL: NCT03840538
Title: Probiotics as a Prophylaxis to Prevent Clinical Manifestations of Oral Candidosis in Patients With Sjogren's Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Kamal Ramadan, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20112012
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probiotic group (Experimental): Probiotic complex capsule taken twice daily for 5weeks
  Interventions: Drug: Probiotic Product - Cap
- Placebo group (Placebo Comparator): Placebo capsule taken twice daily for 5 weeks
  Interventions: Drug: Probiotic Product - Cap

INTERVENTIONS:
Drug: Probiotic Product - Cap — probiotic capsule complex composed of L.acidophilus, L. bulgaricus, Streptococcus thermophilus, and Bifidobacterium bifidus

SUMMARY:
Sjogren's syndrome is an autoimmune chronic disease. It has two forms Primary Sjogren's syndrome charactrized by dry eyes and dry mouth. Secondary Sjogren's syndrome characterized by rheumatoid diseases as rheumatoid arthritis, scleroderma and lupus erythematosus. SS patients are most liable to oral candidiasis , so they need prophylaxis aganist oral candidiasis. Probiotic bacteria are live microorganisms that when administered in adequate amounts confer benefits to health.Probiotics are commonly used as a prophylaxis aganist oral candidosis.

ELIGIBILITY:
Inclusion Criteria:

* primary or scondary Sjogren's syndrome

Exclusion Criteria:

* allergy to milk derivatives previous intake of antifungals

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 5 WEEKS
  Numerical Rating Scale ( NRS)

SECONDARY OUTCOMES:
Candidal load | 5 weeks
  colony forming unit CFU/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Kamal Y, Kandil M, Eissa M, Yousef R, Elsaadany B. Probiotics as a prophylaxis to prevent oral candidiasis in patients with Sjogren's syndrome: a double-blinded, placebo-controlled, randomized trial. Rheumatol Int. 2020 Jun;40(6):873-879. doi: 10.1007/s00296-020-04558-9. Epub 2020 Mar 26. PMID 32219478